CLINICAL TRIAL: NCT00352677
Title: A Phase I, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of INNO-406 in Adult Patients With Imatinib-Resistant or Intolerant Philadelphia Chromosome-Positive (Ph+) Leukemias
Brief Title: Safety and Tolerability Study of INNO-406 to Treat Chronic Myeloid Leukemia or Acute Lymphocytic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CytRx (Industry)
Responsible Party: Michael Dowd, Director, Product Development, Innovive Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INNO-406
Record Dates: First submitted 2006-07-14; First posted 2006-07-17 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Chronic Myeloid Leukemia; Acute Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — bafetinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: INNO-406 — Oral, twice daily self-administration of 10 mg and/or 50 mg tablets

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of INNO-406 in adult patients with imatinib-resistant or intolerant Philadelphia chromosome-positive (Ph+) leukemias.

DETAILED DESCRIPTION:
The purpose of this study is to determine the safety, tolerability and pharmacokinetic profile of INNO-406 when administered as a daily oral agent in adult patients with imatinib-resistant or intolerant Philadelphia chromosome-positive (Ph+) leukemias.

ELIGIBILITY:
Inclusion Criteria:

1. Have a confirmed diagnosis of Ph+ ALL or CML in chronic, accelerated, or blastic phases that are either resistant to or intolerant of imatinib therapy.
2. Be ≥18 years old.
3. Have an Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2.
4. Have an estimated life expectancy of ≥12 weeks.
5. Be male or non-pregnant, non-lactating female. Patients who are fertile must agree to use an effective barrier method of contraception while on therapy and for 90 days following discontinuation of study drug.
6. Have a negative serum or urine pregnancy test within 7 days prior to the first dose of study drug (if patient is a female of childbearing potential).
7. Have acceptable pre-treatment clinical laboratory results.

Exclusion Criteria:

1. Have received chemotherapy ≤1 week from the start of therapy, with the exception of hydroxyurea and corticosteroids.
2. Have received imatinib ≤3 days prior to enrollment or have not recovered from side effects of imatinib therapy.
3. Have impaired cardiac function.
4. Have an active, uncontrolled systemic infection considered opportunistic, life-threatening, or clinically significant at the time of treatment.
5. Have clinically significant acute or chronic liver or renal disease considered unrelated to tumor.
6. Have impaired gastrointestinal function that may significantly alter drug absorption (e.g., uncontrolled vomiting, ulcerative colitis, malabsorption, or small bowel resection).
7. Are pregnant or lactating.
8. Have psychiatric disorder(s) that would interfere with consent, study participation, or follow-up.
9. Have not recovered from acute toxicity of all previous therapy prior to enrollment.
10. Have any other severe concurrent disease and/or uncontrolled medical conditions, which, in the judgment of the investigator, could predispose patients to unacceptable safety risks or compromise compliance with the protocol.
11. Have a history of another primary malignancy that is currently clinically significant or requires active intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose (MTD) and dose limiting toxicity (DLT) of INNO-406 when administered as a single agent to adult patients with imatinib-resistant or intolerant Ph+ leukemias. | One year
To determine the safety profile (including acute and chronic toxicities) and tolerability of INNO-406 in this patient population. | One year

SECONDARY OUTCOMES:
To determine the pharmacokinetic (PK) profile of INNO-406. | One year
To assess BCR-ABL transcript levels and to analyze BCR-ABL mutations. | One year
To assess leukemia response rates in this patient population. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Hagop Kantarjian, M.D., Principal Investigator — University of Texas, MD Anderson Cancer Center, Houston, TX 713-792-7026 hkantarj@mdanderson.org
Locations (6):
- United States (2):
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Texas MD Anderson Cancer Center, Houston, Texas
- Germany (3):
  - Charite University of Medicine, Berlin
  - Johann Wolfgang Goethe Universität, Frankfurt am Main
  - University of Heidelberg Medical Clinic, Mannheim
- Chaim Sheba Medical Center, Tel Litwinsky, Israel